CLINICAL TRIAL: NCT05596812
Title: A Novel Care Pathway in Women With "Low-risk" Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-065
Record Dates: First submitted 2022-07-28; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Risk Stratification Pathway) (Experimental): Those randomized to Intervention (Risk Stratification Pathway) will have their demographic and clinical data entered into the risk stratification screening calculator, and will be assigned to either "Low Risk" (Novel (Low Impact) Care Pathway) or "High Risk" (Routine Care Pathway) groups.
  Women in the Routine Care Pathway group will be followed in the DIP clinic according to routine care protocols and will provide bi-weekly glucometer data.
  Women in the Novel (Low Impact) Care Pathway group will be followed in the New Care Pathway, which will include continuation of lifestyle and dietary modification, continuation of capillary self blood glucose monitoring, and routine prenatal care.
  Interventions: Other: New Care Pathway
- Control (Routine Care) (No Intervention): Those randomized to Control (Routine Care) will continue in-person and virtual visits as per routine care protocols. This group will also provide bi-weekly glucometer data.

INTERVENTIONS:
Other: New Care Pathway — The New Care Pathway will include continuation of lifestyle and dietary modification, self-blood glucose monitoring, and routine prenatal care.
  Arms: Intervention (Risk Stratification Pathway)

SUMMARY:
This study is a randomized controlled trial to study the effect of the use of a risk stratification screening tool for high- and low-risk gestational diabetes mellitus (GDM), and the implementation of a new low-impact care pathway for women with low-risk GDM. The study will measure how well the screening tool and new care pathway are used, and the effect of the new low-impact care pathway on glycemic control, perinatal outcomes (large for gestational age, rate of labor induction, mode of delivery, obstetric anal sphincter injury, neonatal hypoglycemia, neonatal anthropometry) and health resource utilization in women with GDM that are at low-risk of dietary therapy failure.

ELIGIBILITY:
Inclusion Criteria:

* Women able to understand and sign the study consent form
* singleton pregnancy
* planning to give birth to at St. Michael's Hospital
* diagnosed with GDM between 24-32 weeks' gestation based on a positive GCT or GTT result as defined by the Canadian Diabetes Association Clinical Practice Guidelines

Exclusion Criteria:

* Women with preexisting diabetes (Type 1 or 2 diabetes)
* multiple gestation, or a diagnosis of GDM before 24 weeks' or after 32 weeks' gestation
* not continuing care at St. Michael's Hospital after the DIP clinic visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the novel risk stratification screening tool | 2 years
  number of patients screened, recruited, consented and randomized as documented in the study recruitment log

SECONDARY OUTCOMES:
Performance of the GDM risk stratification tool | 2 years
  With regards to identification of women with GDM who maintain euglycemia on lifestyle modification alone in the "Low-risk GDM" group. Sensitivity, specificity, and accuracy will be calculated.
Glycemic control - blood glucose (units) | approximately 9 months (from recruitment at 24-32 weeks gestation to 3-months postpartum)
  mean Fasting Plasma Glucose (FPG) and Post-Prandial Glucose (PPG) in mg/dL
Glycemic control - blood glucose (percent above target) | approximately 9 months (from recruitment at 24-32 weeks gestation to 3-months postpartum)
  percent above target Fasting Plasma Glucose (FPG) and Post-Prandial Glucose (PPG)
Gestational weight gain | approximately 9 months (from recruitment at 24-32 weeks gestation to 3-months postpartum)
  in kilograms (kg)
Development of hypertensive disorders of pregnancy | approximately 9 months (from recruitment at 24-32 weeks gestation to 3-months postpartum)
  documented as recorded from patient charts (Yes/No)
Delivery outcomes - gestational age at delivery | recorded at time of delivery
  measured in weeks
Delivery outcomes - mode of delivery | recorded at time of delivery
  vaginal/caesarean/spontaneous/instrumental/forceps/vacuum/combined
Neonatal outcomes - size for gestational age | recorded at time of delivery
  measured in grams
Neonatal outcomes - Appearance, Pulse, Grimace, Activity, Respiration (APGAR) score | recorded at delivery (at 1 minute and 5 minutes of age)
  Appearance, Pulse, Grimace, Activity, Respiration (APGAR) score is based on a total score of 1 to 10; The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2. A score of 7 or above on the test is considered in good health. A lower score does not mean that the baby is unhealthy, but that the baby may need some immediate medical care, such as suctioning of the airways or oxygen to help him or her breathe better.
Health service outcomes - health resource utilization | 2 years
  total number of care encounters (categorized by department - endocrine, obstetric)
Health service outcomes - Short-form Patient Satisfaction Questionnaire (PSQ-18) | 2 years; administered to each participant at 6-weeks postpartum
  Short-form Patient Satisfaction Questionnaire (PSQ-18); responses to items are measured on a 5-point Likert scale (1 = Strongly Agree, 5 = Strongly Disagree). Minimum score is 18, maximum score is 90. Higher scores indicate satisfaction with medical care.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital (Unity Health Toronto), Toronto, Ontario, Canada